CLINICAL TRIAL: NCT05270538
Title: Cardiorespiratory and Acid-basic Imbalance Caused by Use of Face Mask, During Physical Exercices
Brief Title: Cardiorespiratory and Acid-basic Imbalance Caused by Use of Mask
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Vale do Sapucai (Other)
Responsible Party: Principal Investigator, José Dias da Silva Neto, Phd, Universidade do Vale do Sapucai
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 5.026.897
Record Dates: First submitted 2022-02-15; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Acid-Base Imbalance; Respiration Disorders
Keywords: Masks; Acid-Base Imbalance; physiology
MeSH Terms: conditions — Acid-Base Imbalance; Respiration Disorders

STUDY DESIGN:
Intervention Model Description: Of the 57 participants, 26 are allocated as G1 (46.5%) and 31 as G2 (53.5%) After the collection of blood gases and cardiovascular parameters- Systolic Blood Pressure, Diastolic Blood Pressure, Heart Rate and O2 Saturation - before and after physical exercise, all participants answered a socio-demographic questionnaire informing their weight, height and gender, in addition to completing the Informed Consent Form on the experiment
Masking Description: Control group (G1) and study group (G2) were defined from the use of random sampling software that gave numbers to each participant, distributing them between the two groups - participants who removed odd numbers were assigned to G1 while participants who removed even numbers to G2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- comparison of clinical and gasometric parameters between the study group and the control group (Active Comparator): To carry out the study, we defined a control group and a study group distributing them between the two groups. The control group will perform the exercise, without using a mask, while the study group will perform the exercise using Masks Zero Mask Sewing Virus Bac-Off Lupo® for the duration of the exercise.
  The exercise consisted of 15 minutes of treadmill without inclination interspersing every 2 minutes at speeds 10 Km/h and 12 Km/h, being by definition of a dynamic aerobic exercise of intensity 4 of 5 in the Borg scale- classification of the intensity of physical exercise. Physical activity was performed in water deprivation and fasting at least 30 minutes before the start of activated.
  Interventions: Device: Mask Zero Seam Virus Bac-Off Lupo® 98% Polyamide and 2% Elastane

INTERVENTIONS:
Device: Mask Zero Seam Virus Bac-Off Lupo® 98% Polyamide and 2% Elastane — The 26 participants allocated as G2 had to perform the physical exercise using the Zero Sewing Virus Bac-Off Virus® 98% Polyamide and 2% Elastane, in order to totally seal the nose and mouth.

SUMMARY:
The study aims to evaluate whether the use of polypropylene and elastane Lupo ® masks can be considered as a significant causal agent in cases of respiratory and acid-base imbalances. For this, gas parameters such as lactate, bicarbonate, Sat02, pH, Sat02, P02 and PC02 of people before and after the practice of aerobic physical exercises will be measured. The control group will perform the exercise without wearing a mask and the study group will perform the exercise using a mask.

DETAILED DESCRIPTION:
The experimental phase was carried out at the Armação Atlética academy accredited by the Medical School of Pouso Alegre, following all sanitary recommendations in relation to covid-19.

The aerobic exercise performed by the participants consisted of 15 minutes of running on the treadmill without inclination, interspersing the speeds 10 km/h and 12km/h.

The evaluated clinical parameters of blood pressure, heart rate, pulse , O2 saturation and biochemical analyses of lactate, (partial oxygen pressure) PO2, (partial pressure of CO2 (carbon dioxide) PC02,(hydrogenic potential) pH ,- were collected just before exercise and shortly after that - with maximum interval between measurements of 2 minutes- through physical examination of the cardiovascular apparatus using littmann classic stetoscope iii®,Multilaser® sphygmomanometer and digital oximeter; and arterial blood collection for blood gas analysis.

The blood gas parameters were obtained before and after exercise from blood sample collection by arterial puncture of the Radial Artery performed by the nurses responsible for the blood gas service of the Samuel Libânio Clinic hospital in order to avoid errors regarding the technique. After collection, the samples were kept in a heparinized container and under cooling in an appropriate thermal box and were sent within 20 minutes to the laboratory to be analyzed by blood gas analysis.Such measures avoided the formation of microclots in the samples and the dissipation of blood gases to be analyzed as Co2 and O2 thus bypassing such possible random bias. The blood gas samples obtained were sent to the Hcsl Clinical Analysis laboratory where they underwent gas run in werfen's GEM Premier 3500® apparatus.

To perform the study, we defined a control group and study group based on the use of random sampling software that gave numbers to each participant, distributing them between the two groups. The control group will perform the exercise, without using a mask, while the study group will perform the exercise using Masks Zero Mask Sewing Virus Bac-Off Lupo® for the duration of the exercise.The specific use of this trademark mask made of 98% Polyamide and 2% Elastane ensures that there will be no variations within the study group regarding the composition of the mask, which could result in variable degrees of seals and, therefore, confounding bias to the study.

As an additional safety measure, especially for participants who have to perform the exercise without mask, since they can reinfect themselves, mobile transparent polymer plates for both groups will be temporarily installed around the treadmill. The appliance will be sanitized after each participant used it, with alcohol 70.

After performing the exercise, participants must complete the socio-demographic form sent via Forms in order to characterize such group regarding gender, weight age of participants.

The data acquired through the experiment received static treatments such as a. Classificationtest Signed by Wilcoxon by the statistician of the University of Vale do Sapucaí- Univás).

ELIGIBILITY:
Inclusion Criteria:

* Healthy medical students who practice physical activity regularly, at least 3 times a week.

Exclusion Criteria:

* people who do not accept to participate in the study, refusing to sign the free and informed consent form.
* Sedentary people
* people with major cardiorespiratory diseases or comorbidity
* people tested positive for Covid-19 or other respiratory-infectious diseases in less that 15 days

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2022-01-12 (Actual)

PRIMARY OUTCOMES:
variation of lactate | This variation of blood parameter was obtained through the blood gas analysis to which the participants were submitted just before the beginning of the physical exercise - with a maximum time interval of 2 minutes- and later comparing these
  arterial puncture for blood gas analysis
variation of pH | This variation of blood parameter was obtained through the blood gas analysis to which the participants were submitted just before the beginning of the physical exercise - with a maximum time interval of 2 minutes- and later comparing these
  arterial puncture for blood gas analysis
variation of P02 | This variation of blood parameter was obtained through the blood gas analysis to which the participants were submitted just before the beginning of the physical exercise - with a maximum time interval of 2 minutes- and later comparing these
  arterial puncture for blood gas analysis
variation of PC02 | This variation of blood parameter was obtained through the blood gas analysis to which the participants were submitted just before the beginning of the physical exercise - with a maximum time interval of 2 minutes- and later comparing these
  arterial puncture for blood gas analysis
variation of Sat02 | This variation of blood parameter was obtained through the blood gas analysis to which the participants were submitted just before the beginning of the physical exercise - with a maximum time interval of 2 minutes- and later comparing these
  arterial puncture for blood gas analysis
variation of bicarbonate | This variation of blood parameter was obtained through the blood gas analysis to which the participants were submitted just before the beginning of the physical exercise - with a maximum time interval of 2 minutes- and later comparing these
  arterial puncture for blood gas analysis
heart rate (bpm) | This variation of blood parameter was obtained through the blood gas analysis to which the participants were submitted just before the beginning of the physical exercise - with a maximum time interval of 2 minutes- and later comparing these
  physical examination of the cardiovascular system
blood pressure | This variation of blood parameter was obtained through the blood gas analysis to which the participants were submitted just before the beginning of the physical exercise - with a maximum time interval of 2 minutes- and later comparing these
  physical examination of the cardiovascular system

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Brandão, PhD, Principal Investigator — Universidade do Vale do Sapucai
Locations (2):
- Brazil (2):
  - Univas, Pouso Alegre, Minas Gerais
  - Univás, Pouso Alegre, Minas Gerais

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brum PC, Da Silva GJ, Moreira ED, Ida F, Negrao CE, Krieger EM. Exercise training increases baroreceptor gain sensitivity in normal and hypertensive rats. Hypertension. 2000 Dec;36(6):1018-22. doi: 10.1161/01.hyp.36.6.1018. PMID 11116118
- [Background] Gava NS, Veras-Silva AS, Negrao CE, Krieger EM. Low-intensity exercise training attenuates cardiac beta-adrenergic tone during exercise in spontaneously hypertensive rats. Hypertension. 1995 Dec;26(6 Pt 2):1129-33. doi: 10.1161/01.hyp.26.6.1129. PMID 7498982
- [Background] Negrao CE, Moreira ED, Brum PC, Denadai ML, Krieger EM. Vagal and sympathetic control of heart rate during exercise by sedentary and exercise-trained rats. Braz J Med Biol Res. 1992;25(10):1045-52. PMID 1342828
- [Background] Medeiros A, Oliveira EM, Gianolla R, Casarini DE, Negrao CE, Brum PC. Swimming training increases cardiac vagal activity and induces cardiac hypertrophy in rats. Braz J Med Biol Res. 2004 Dec;37(12):1909-17. doi: 10.1590/s0100-879x2004001200018. Epub 2004 Nov 17. PMID 15558199
- [Background] Seccareccia F, Menotti A. Physical activity, physical fitness and mortality in a sample of middle aged men followed-up 25 years. J Sports Med Phys Fitness. 1992 Jun;32(2):206-13. PMID 1434592
- [Background] Forjaz CL, Tinucci T, Ortega KC, Santaella DF, Mion D Jr, Negrao CE. Factors affecting post-exercise hypotension in normotensive and hypertensive humans. Blood Press Monit. 2000 Oct-Dec;5(5-6):255-62. doi: 10.1097/00126097-200010000-00002. PMID 11153048
- [Background] Forjaz CL, Cardoso CG Jr, Rezk CC, Santaella DF, Tinucci T. Postexercise hypotension and hemodynamics: the role of exercise intensity. J Sports Med Phys Fitness. 2004 Mar;44(1):54-62. PMID 15181391
- [Background] Porcari JP, Probst L, Forrester K, Doberstein S, Foster C, Cress ML, Schmidt K. Effect of Wearing the Elevation Training Mask on Aerobic Capacity, Lung Function, and Hematological Variables. J Sports Sci Med. 2016 May 23;15(2):379-86. eCollection 2016 Jun. PMID 27274679
- [Background] Reis JF, Millet GP, Malatesta D, Roels B, Borrani F, Vleck VE, Alves FB. Are oxygen uptake kinetics modified when using a respiratory snorkel? Int J Sports Physiol Perform. 2010 Sep;5(3):292-300. doi: 10.1123/ijspp.5.3.292. PMID 20861520
- [Background] Ngomane AY, Fernandes B, Guimaraes GV, Ciolac EG. Hypotensive Effect of Heated Water-based Exercise in Older Individuals with Hypertension. Int J Sports Med. 2019 Apr;40(4):283-291. doi: 10.1055/a-0828-8017. Epub 2019 Feb 21. PMID 30791079
- [Background] Teodoro CL, Gaspari AF, Berton R, Barbieri JF, Silva M, A A Castano L, Guimaraes P, Moraes AC. Familiarization With Airflow-Restriction Mask During Resistance Exercise: Effect on Tolerance and Total Volume. J Strength Cond Res. 2019 Jul;33(7):1762-1765. doi: 10.1519/JSC.0000000000002828. PMID 30204655
- [Background] Kellum JA. Disorders of acid-base balance. Crit Care Med. 2007 Nov;35(11):2630-6. doi: 10.1097/01.CCM.0000286399.21008.64. PMID 17893626
- [Background] MacIntyre CR, Zhang Y, Chughtai AA, Seale H, Zhang D, Chu Y, Zhang H, Rahman B, Wang Q. Cluster randomised controlled trial to examine medical mask use as source control for people with respiratory illness. BMJ Open. 2016 Dec 30;6(12):e012330. doi: 10.1136/bmjopen-2016-012330. PMID 28039289
- [Background] Eikenberry SE, Mancuso M, Iboi E, Phan T, Eikenberry K, Kuang Y, Kostelich E, Gumel AB. To mask or not to mask: Modeling the potential for face mask use by the general public to curtail the COVID-19 pandemic. Infect Dis Model. 2020 Apr 21;5:293-308. doi: 10.1016/j.idm.2020.04.001. eCollection 2020. PMID 32355904